CLINICAL TRIAL: NCT02318914
Title: A 2-Year, Open-Label, Safety Extension Study of Gevokizumab in Patients With Pyoderma Gangrenosum
Brief Title: A 2-Year, Open-Label, Safety Extension Study of Gevokizumab in Subjects With Pyoderma Gangrenosum
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X052171
Record Dates: First submitted 2014-12-08; First posted 2014-12-17 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Pyoderma Gangrenosum
Keywords: Pyoderma Gangrenosum; Classic Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — gevokizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gevokizumab (Experimental): Solution for subcutaneous injection
  Interventions: Drug: gevokizumab

INTERVENTIONS:
Drug: gevokizumab

SUMMARY:
The study will evaluate the long-term safety of gevokizumab in treating active PG ulcers

ELIGIBILITY:
Inclusion Criteria:

* Individuals who participated in a previous study of gevokizumab in PG
* A clinical diagnosis of classic pyoderma gangrenosum
* Contraceptive measures adequate to prevent pregnancy during the study

Exclusion Criteria:

* Clinical evidence of acutely infected pyoderma gangrenosum
* History of allergic or anaphylactic reactions to monoclonal antibodies
* History of recurrent or chronic systemic infections
* Female subjects who are pregnant, planning to become pregnant, have recently delivered, or are breast-feeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment-emergent adverse events; | Up to 2 years
Changes from baseline vital signs, physical examination results, and laboratory test results | Up to 2 years
Changes from baseline concomitant medications use | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (40):
- United States (31):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Oceanside, California
  - San Diego, California
  - Farmington, Connecticut
  - Coral Gables, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Henderson, Nevada
  - Lebanon, New Hampshire
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Lubbock, Texas
  - Salt Lake City, Utah
- Australia (7):
  - Benowa, Queensland
  - Woolloongabba, Queensland
  - Parkville, Victoria
  - Fremantle
  - St Leonards
  - Sydney
  - Westmead
- Canada (2):
  - Markham, Ontario
  - Richmond Hill, Ontario